CLINICAL TRIAL: NCT02299804
Title: A Multicenter, Double-Blind, Phase Ⅱ Clinical Trial To Evaluate Efficacy And Safety Of Levophencynonate Hydrochloride In Patient With Vertigo Caused By Posterior Circulation Infarction
Brief Title: A Clinical Trial To Evaluate Efficacy And Safety Of Levophencynonate Hydrochloride In Patient With Vertigo
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sihuan Pharmaceutical Holdings Group Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LEVO-PCIV-2001
Record Dates: First submitted 2014-10-09; First posted 2014-11-24 (Estimated); Last update posted 2016-04-15 (Estimated); Status verified 2016-04

CONDITIONS: Vertigo
MeSH Terms: conditions — Vertigo

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- High dose arm (Experimental): Have included the Levophencynonate Hydrochloric 1.5mg bid.
  Interventions: Drug: Levophencynonate Hydrochloric
- Low dose arm (Experimental): Have included the Levophencynonate Hydrochloric 1.0mg bid.
  Interventions: Drug: Levophencynonate Hydrochloric
- Placebo arm (Placebo Comparator): Have no any active component
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Levophencynonate Hydrochloric — this drug is M receptor inhibitor
  Arms: High dose arm; Low dose arm
Drug: Placebo — No active ingredient
  Arms: Placebo arm

SUMMARY:
A Multicenter, Double-Blind, Placebo Controlled, Phase Ⅱa clinical trial to enroll 120 patients with Vertigo Caused By Posterior Circulation Infarction during 7 days, then to evaluate the efficacy of different dose of Levophencynonate Hydrochloric, and provide the effective dosage for phase IIb clinical study, to study the safety of Levophencynonate Hydrochloric.

DETAILED DESCRIPTION:
This study will conduct in 15 sites to enrolled 120 patients with vertigo under 7 days treatment and 7 days follow-up. The study includes three arms: high dose, low dose and placebo control.To observe the efficacy by change of vertigo severity and duration,and safety by vital sign,adverse event,etc.

ELIGIBILITY:
Inclusion Criteria:

1. At the age more than 18 years old male or female;
2. Patients with vertigo caused by Posterior Circulation Infarction.
3. Patients diagnosed Posterior Circulation Infarction based on the criteria of Posterior Circulation Ischemia of America;
4. Meet the diagnose criteria of vertigo: Visual Motion (External Vertigo), or Rotation, Swing, Lift and Tilt Sensation (Internal Vertigo);
5. Ability to sign the statements of informed consent;

Exclusion Criteria:

1. Female patients having Pregnant, Lactating or Birth plan recently;
2. Non-posterior circulation infarction patients;
3. Vertigo caused by any other diseases;
4. Long-term alcohol abuse, or drug abuse;
5. Been in critical condition, difficult to make a precise evaluation of efficacy and safety of new drugs;
6. History of allergies on Levophencynonate Hydrochloric or these compositions;
7. Participation in another clinical trial in three months;
8. Investigator thought that should be excluded due to other reason;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2014-01; Primary Completion 2015-05 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
The duration of vertigo | up to 7 days
  The Software Statistical Analysis System (SAS) will be used to deal with 98 subjects' data in the trial. The descriptive statistics will be presented for all efficacy and safety variables. All of questionnaire will be resolved by investigator detailed. Hypothesis test results of effectiveness provide evidence as reference.

SECONDARY OUTCOMES:
Vertigo severity improved（VAS score） | up to 7 days
  The Software Statistical Analysis System (SAS) will be used to deal with the 98 patients' data in the trial. The descriptive statistics will be presented for all efficacy and safety variables. All of questionnaires will be resolved by investigator.Hypothesis test results of effectiveness provide evidence as reference.
Nerve function improved（NIHSS/MRS score） | up to 7 days
  The Software Statistical Analysis System (SAS) will be used to deal with the 98 patients' data in the trial. The descriptive statistics will be presented for all efficacy and safety variables. All of questionnaires will be resolved by investigator.Hypothesis test results of effectiveness provide evidence as reference.

CONTACTS AND LOCATIONS:
Overall Officials: Yansheng Li, PHD, Principal Investigator — RenJi Hospital
Locations (1):
- Renji Hospital Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No